CLINICAL TRIAL: NCT04769414
Title: A Phase II Trial of Flouro-Gem as a First Line Treatment of Metastatic Adenocarcinoma of the Pancreas (GEFLUPAN)
Brief Title: Flouro-Gem in Adenocarcinoma of the Pancreas (GEFLUPAN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed Sohaib, Lecturer of Clinical oncology, Menoufia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 352
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Cancer of Pancreas; Chemotherapy Effect; Metastatic Pancreatic Cancer
Keywords: pancreas; cancer; adenocarcinoma; metastatic; gemcitabine; flourouracil; chemotherapy; first line
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Adenocarcinoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Experimental): Participants will receive the test protocol Gem-5FU on biweekly basis for 6 months with interim evaluation
  Doses as follows:
  Gemcitabine 1000 mg/m2, infusion over 30 min, D1, D15 Leucovorin 400 mg/m2 infusion over 30 min , D1, D15 5FU 400 mg/m2 I.V. shot D1, D15 5FU 2000 mg/m2 infusion over 46 hours D1 , D15
  Interventions: Drug: Gemcitabine fluorouracil

INTERVENTIONS:
Drug: Gemcitabine fluorouracil — chemotherapy protocol given as:
  * Gemcitabine 1000mg/m2 IV short infusion
  * Leucovorin 400 mg/m2 IV short infusion
  * Flourouracil 400 mg/m2 direct IV shot
  * Flourouracil 2000 mg/m2 contineous infusion over 46 hours
  The whole regimen will be repeated bi-weekly

SUMMARY:
In this study, the investigators designed a treatment regimen including the most active agents in pancreatic cancer which are gemcitabine and fluorouracil to be tested as a first line treatment. This regimen is expected to be less toxic than FOLFIRINOX and aiming at better outcomes.

DETAILED DESCRIPTION:
Metastatic cancer pancreas has been a challenge for oncologists over the years. It is a disease of limited survival and a very poor response to treatment. The median overall survival at five years is expected to be between 4-6% only. Adenocarcinoma is the most common type of pancreatic cancer. It is the tenth most common adult solid malignancy. Most of the new therapeutic modalities has proven to be non-beneficial in this disease including targeted and immunotherapy.

For many years, the first line of treatment for pancreatic cancer was gemcitabine either alone or in combinations. Recently, FOLFIRINOX has become the standard of care due to its overall survival benefit. However, it is a small benefit on the expense of great toxicity.

Patients with metastatic cancer pancreas are recruited to receive the test regimen. Baseline evaluation will be done either by CT scan or PET/CT. re-evaluation will be repeated after 3 months of treatment and at end of 6 months

ELIGIBILITY:
Inclusion Criteria:

* Histopathological evidence of adenocarcinoma of the pancreas
* Radiological proof of metastatic disease as defined by AJCC

Exclusion Criteria:

* patients with poor performance status (ECOG 4)
* patients with organ dysfunction defined as: creatinine more than 1.6 mg/dl or bilirubin more than 3 mg/dl
* patients with end stage renal disease who are under regular dialysis
* other histologies of pancreatic cancer
* irresectable pancreatic cancer if not metatatic

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-07-09 (Actual); Study Completion 2022-07-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 months from enrollment
  describes according to RECIST criteria

SECONDARY OUTCOMES:
Adverse events (AE) | 6 months from chemotherapy
  Describes according to CTCAE
Progression free survival (PFS) | One year from start of enrollment
  The time interval between the date of metastasis to the date of next disease progression
Overall survival (OS) | One year from start of enrollment
  The time interval between the date of diagnosis till the date of death

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Faculty of medicine, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared with other investigators upon personal contact with the PI of the study and after publishing the primary results. The investigators of this study are to be submitted as co-investigators in any other studies using the data of this study.
Supporting Information: Study Protocol, SAP
Time Frame: After publishing the primary results of the study, expected to be by January 2023

REFERENCES:
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347